CLINICAL TRIAL: NCT03136653
Title: A Phase 2 Open-label, Single-arm, Multicenter Trial of MP0250 Plus Bortezomib + Dexamethasone in Patients With Refractory and Relapsed Multiple Myeloma
Brief Title: A Phase 2 Trial of MP0250 Plus Bortezomib + Dexamethasone in Patients With Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Molecular Partners AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP0250-CP201; 2016-002771-10 (EudraCT Number)
Record Dates: First submitted 2017-04-18; First posted 2017-05-02 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Multiple Myeloma in Relapse
Keywords: DARPin; MP0250; VEGF; HGF; RRMM
MeSH Terms: interventions — MP0250

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm Study MP0250 plus BOR + DEX (Experimental): Single arm study of MP0250 plus bortezomib + dexamethasone
  Interventions: Biological: MP0250 plus BOR+DEX

INTERVENTIONS:
Biological: MP0250 plus BOR+DEX — 6 mg/kg or 8 mg/kg or 12 mg/kg of MP0250, IV (in the vein,) on day 1 of each 21 day cycle. Bortezomib and Dexamethasone according to label.
  Number of Cycles: until progression or unacceptable toxicity develops.

SUMMARY:
The purpose of this study is to assess the efficacy, safety, tolerability, pharmacokinetics (PK), immunogenicity and efficacy of MP0250 in combination with bortezomib + dexamethasone in patients with refractory and relapsed multiple myeloma (RRMM).

MP0250 is a multi-DARPin® drug candidate with three specificities, able to simultaneously neutralize the activities of vascular endothelial growth factor (VEGF) and hepatocyte growth factor (HGF) and also to bind to human serum albumin (HSA) to give an increased plasma half-life and potentially enhanced tumor penetration.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with MM who have received:

   * Part 1 ≥2 lines of therapy (including bortezomib and an IMiD) and have shown no response (i.e. stable disease) to, have progressed on the most recent treatment or have progressed within 60 days of the most recent therapy
   * Part 2 ≥2 lines of prior therapy that included a proteasome inhibitor (bortezomib, carfilzomib or both) and an IMiD (thalidomide, lenalidomide and/or pomalidomide) either alone or in combination and a response no better than SD lasting at least 4 months on a bortezomib- or carfilzomib-based regimen as last line of therapy or progression on treatment or within 60 days of stopping a bortezomib- or carfilzomib-based regimen as last line of therapy. Note: For transplant-eligible patients enrolled to Part 1 or Part 2, induction plus conditioning chemotherapy/ASCT +/- maintenance therapy constitute one regimen.
2. Presence of a measurable disease with at least one of the following criteria:

   * Serum M protein ≥0.5 g/dL, or
   * Urine M protein ≥200 mg/24 h, or
   * Involved serum free light chain (FLC) levels >100 mg/L and abnormal kappa/lambda (κ/λ) ratio in patients without detectable serum or urine M protein, or
   * For patients with immunoglobulin A (IgA) myeloma whose disease can only be reliably measured by quantitative immunoglobulin measurement, a serum IgA level ≥0.5g/dL.
3. Eastern Cooperative Oncology Group (ECOG) performance status (0 to 1)
4. Life expectancy >3 months
5. Adequate hepatic function at Screening, with aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <3x ULN and total bilirubin <2 x upper limit of normal (ULN). For patients with Gilbert's syndrome (Gilbert-Meulengracht syndrome), higher bilirubin of 5 x ULN is acceptable
6. Absolute neutrophil count (ANC) ≥1000/mm3 at Screening. Screening ANC must be independent of growth factor support for ≥1 week
7. Hemoglobin ≥8.0 g/dL at Screening. Use of erythropoietic stimulating factors and red blood cell (RBC) transfusions per institutional guidelines is allowed, however most recent RBC transfusion must not have been done within 7 days prior to obtaining screening hemoglobin
8. Platelet count ≥50 000/mm3 at Screening. Patients must not have received platelet transfusions for at least 1 week prior to obtaining the screening platelet count
9. Calculated or measured creatinine clearance (CrCl) of ≥ 45 mL/min at Screening based on the Cockcroft and Gault formula
10. Serum albumin concentration ≥ 25 g/L. Note: Patients with lower levels of serum albumin at baseline may receive albumin supplementation to comply with this criterion
11. Males and females ≥18 years of age
12. Male Participants: A male participant must agree to use a highly effective contraception
13. Female Participants: A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

    1. Not a woman of childbearing potential (WOCBP) OR
    2. A WOCBP who agrees to follow contraceptive guidance from the Screening visit, during the treatment period and for at least 3 months after the last dose of study treatment
14. Capable of giving signed informed consent

Exclusion Criteria:

1. Patients with the following diseases:

   * Monoclonal gammopathy of undetermined significance (MGUS) of non- immunoglobulin (Ig)M and IgM subtypes,
   * Light chain MGUS,
   * Solitary plasmacytoma (alone or with minimal marrow involvement),
   * Systemic Ig light chain amyloidosis,
   * Waldenstrom's Macroglobulinemia,
   * Myelodysplastic syndrome,
   * Plasma cell leukemia defined as a plasma cell count >2000/mm3
   * Polyneuropathy, organomegaly endocrinopathy, monoclonal protein, and skin changes (POEMS) syndrome
2. Peripheral neuropathy Grade 2 or higher at Screening or patients with a history of Grade 3/4 neuropathy or Grade 2 with pain
3. Prior or concurrent malignancy, except for: Adequately treated basal cell or squamous cell skin cancer, carcinoma in-situ of the cervix or breast or very low and low risk prostate cancer in active surveillance or any other cancer from which the patient has been disease-free for >5 years
4. Active congestive heart failure (New York Heart Association [NYHA] Class III to IV), symptomatic cardiac ischemia, or conduction abnormalities uncontrolled by conventional intervention. Myocardial infarction within 6 months prior to screening
5. Uncontrolled hypertension (defined as systolic blood pressure (SBP) >150 mm Hg diastolic blood pressure (DBP) >100 mm Hg despite antihypertensive medication)
6. Stroke, or transient ischemic attack within 6 months of Screening, clinically significant bleeding and vascular disease
7. Abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
8. Significant concurrent, uncontrolled medical condition including, but not limited to, severe wound healing complication, renal (except related to MM), hepatic, hematological except MM, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease
9. Acute active infection requiring systemic antibiotics, antiviral (except antiviral therapy directed at hepatitis B) or antifungal agents within 14 days prior to screening
10. Clinical signs of or documented leptomeningeal or cerebral involvement of MM
11. Treatment with ixazomib as last line of therapy in Part 2
12. Therapy with approved or investigational anticancer therapeutics within 21 days (or in the case of nitrosureas, within 6 weeks) prior to treatment (except anti-myeloma treatment with a carfilzomib- or bortezomib-based regimen in Part 2) Note: Patients must have recovered from pre-existing, treatment-related adverse events to Grade 1 or lower
13. Autologous stem cell transplantation (ASCT) within 12 weeks before the date of enrollment
14. Prior allogeneic stem cell transplantation with active graft-versus-host-disease
15. Major surgery within 21 days prior to Screening
16. Immunotherapy within 21 days prior to Screening
17. Newly initiated therapy with bisphosphonate or RANKL (within two months prior to Screening). Patients on stable regimen with bisphosphonate or receptor activator of nuclear kappa-B ligand (RANKL)-inhibitor therapy over 2 months can continue these treatments at the same dose. No new therapy with bisphosphonate/RANKL inhibitor is allowed during the study
18. Radiation therapy within 2 months of Cycle 1, Day 1 is not permitted Except for local low-dose, palliative radiation to bone lesions for pain control.
19. Patients who have received treatment with any non-marketed product within 21 days prior to treatment start
20. Current participation in any other interventional clinical study
21. Patients known or suspected of not being able to comply with a study protocol (e.g. due to alcoholism, drug dependency or psychological disorder)
22. Known infection with human immunodeficiency virus or serologic status reflecting active hepatitis B or hepatitis C virus infection as follows:

    * Not receiving or not responding to anti-viral therapy.
    * HCV RNA detected
23. Patients with contraindication to dexamethasone or bortezomib according to the applicable local product label
24. Known hypersensitivity to components of the investigational product, for example, histidine buffer or the Tween diluent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2020-10-12 (Actual); Study Completion 2021-01-13 (Actual)

PRIMARY OUTCOMES:
Part 1: Overall Response Rate (ORR) | 24 months
  Defined as the number of participants achieving a complete response (CR), very good partial response (VGPR), or partial response (PR) during treatment with MP0250 plus bortezomib+dexamethasone determined by the Investigator in part 1.
Part 2: ORR | 24 months
  Defined as the number of participants achieving a confirmed, stringent complete response (sCR), very good partial response (VGPR), or partial response (PR) during treatment with MP0250 plus bortezomib+dexamethasone determined by the Investigator in part 2.

SECONDARY OUTCOMES:
Number of Participants Who Experienced One or More Treatment-Emergent Adverse Events | 24 months
Number of Participants who Experienced One or More Treatment-Emergent SAEs | 24 months
Number of Participants Who Experienced One or More Common Terminology Criteria for Adverse Events (CTCAE) Grade ≥ 3 Adverse Events | 24 months
Number of Participants with a Clinical Significant Change from Baseline in Laboratory Results | 24 months
Number of Participants with a Clinically Significant Change from Baseline in Vital Signs | 24 months
Number of Participants with a Clinically Significant Change from Baseline in Electrocardiogram (ECG) Results | 24 months
Number of Participants with a Positive Anti-drug Antibody (ADA) Result | 24 months
Titer of Anti-drug Antibodies (ADA) | 24 months
Time Course of Anti-drug Antibodies | 24 months
Duration of Response (DOR) | 24 months
  DOR is defined as the duration from first observation of partial response (PR) or better until disease progression, or death from myeloma.
Progression Free Survival (PFS) | 24 months
  PFS is determined as the time from first study treatment until progression or death from myeloma.

CONTACTS AND LOCATIONS:
Locations (24):
- Austria (2):
  - Hanusch Krankenhaus Wiener Gebietskrankenkasse, Vienna, Vienna
  - Landeskliniken Salzburg Saint Johanns-Spital, Salzburg
- Czechia (2):
  - Fakultní Nemocnice Brno, Brno, Jihormoravsky Krav
  - Fakultní Nemocnice Ostrava, Ostrava - Poruba, Severomoravsky KRAJ
- Denmark (2):
  - Odense University Hospital, Odense C
  - Vejle Sygehus, Vejle
- Germany (7):
  - Asklepios Klinik Altona, Altona, Hamburg
  - Universitätsklinikum Dresden, Dresden, Saxony
  - Universitaetsklinikum Essen, Essen
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsklinikum Münster, Münster
  - Universitätsklinikum Würzburg, Würzburg
- Italy (5):
  - Azienda Ospedaliera Policlinico di Bari, Bari
  - Azienda Ospedaliero Universitaria di Bologna Policlinico Sant'Orsola-Malpighi, Bologna
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Torino
- Poland (6):
  - Samodzielny Publiczny Zakład Opieki Zdrowotnej Zespół Szpitali Miejskich, Chorzów, Silesian Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Centrum Onkologii Ziemi Lubelskiej, Lublin
  - Szpital Wojewódzki w Opolu, Opole
  - Instytut Hematologii i Transfuzjologii, Warsaw

IPD SHARING:
Plan to Share IPD: No